CLINICAL TRIAL: NCT01936545
Title: The Impact of Different Anesthetic Methods on Ischemia Reperfusion Injury Following Liver Transplantation
Brief Title: Anesthetic Methods and Liver Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201003116M
Record Dates: First submitted 2013-08-27; First posted 2013-09-06 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Acute Lung Injury
Keywords: Liver transplantation, reactive oxygen species, antioxidant
MeSH Terms: conditions — Acute Lung Injury | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- propofol (Experimental): The anesthesia was maintained with propofol during liver transplantation.
  Interventions: Drug: propofol during liver transplantation.
- Desflurane (Active Comparator): The anesthesia was maintained with desflurane during liver transplantation.
  Interventions: Drug: Desflurane during liver transplantation.

INTERVENTIONS:
Drug: propofol during liver transplantation. — The anesthesia was maintained with propofol during liver transplantation.
  Other Names: propofol
  Arms: propofol
Drug: Desflurane during liver transplantation. — The anesthesia was maintained with desflurane during liver transplantation.
  Other Names: Desflurane
  Arms: Desflurane

SUMMARY:
Postoperative pulmonary complications are not uncommon after liver transplantation. They can not only prolong the stay in intensive care unit and in hospital but also increase the morbidity and mortality rate. The underlying mechanisms are multifactorial, however, oxidative stress following hepatic ischemia reperfusion and the ensuing pulmonary leukocyte infiltration play an important part in the pulmonary complications. Various drugs and methods such as ischemic preconditioning have been used to lessen the production of oxidative free radicals following hepatic ischemia reperfusion. The choice of different anesthetic agents could aslo change the degree of production of oxygen species and antioxidant capacity during the operation.

Volatile and intravenous anesthetic agents can decrease oxidative injuries through different mechanisms, however, which is better in preventing the pulmonary leukocyte infiltration is still unknown.

We attempt the compare the oxidative stress and cytokine level in liver transplant recipients under desflurane or propofol anesthesia to evaluate which kind of anesthetic agent is better in this kind of surgery.

DETAILED DESCRIPTION:
The occurrence of postoperative pulmonary complications after hepatic reperfusion, such as in patients undergoing liver transplantation, is a major concern in the intensive care unit. Not only neutrophil infiltration, but also oxidative injuries, have been demonstrated after intra-operative hepatic ischemia/reperfusion (I/R) management. Previous studies have shown that reactive oxygen species (ROS) paly a major role in the ensuing damage, although I/R-induced remote organ injury is a complex and multifactorial process. Methods to reduce ROS generation, such as ischemic preconditioning, attenuate both liver and lung damage after hepatic I/R. Considering the intra-operative ROS production occurs after hepatic reperfusion , the choice of anesthetics may alter the magnitude of ROS production and the antioxidant capacity.

Volatile and non-volatile anesthetics can exert their antioxidant capacity through different mechanisms. Propofol (2,6-diisopropylphenol) has been reported to provide antioxidant capacity by scavenging free radicals. However, volatile anesthetics such as isoflurane, desflurane or sevoflurane can reduce the oxidative damage through anesthetic preconditioning. Several animal studies demonstrate that volatile anesthetics offer more protection against ischemia-reperfusion injury than intravenous anesthetics. On the contrary, intravenous anesthetics may be more protective against sepsis-induced hepatic injury than volatile anesthetics. However, there are few investigations concerning the effects of different anesthetics on remote pulmonary injuries in clinical settings.

In this study, propofol and desflurane will be used for the maintenance of anesthesia during liver transplantation. The heart function, respiratory function, liver function, kidney function, the oxidative injuries and inflammatory mediators will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* End stage liver disease scheduled for liver transplantation in National Taiwan University Hospital

Exclusion Criteria:

* Pre-existing pulmonary disease
* coma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2011-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change of cardiac output perioperatively | one week
  Cardiac output(l/min) was measured by thermodilution method perioperatively.

SECONDARY OUTCOMES:
lung injury score | one week
  PaO2/FiO2(Arterial oxygen tension/fraction of inspired oxygen)

OTHER OUTCOMES:
Reactive oxygen species | one week
  Reactive oxygen species measured by chemiluminescence method

CONTACTS AND LOCATIONS:
Overall Officials: Kuang Cheng Chan, M.D., Principal Investigator — Department of Anesthesiology, NTUH, Taipei, Taiwan
Locations (1):
- Department of Anesthesiology, NTUH, Taipei, Taiwan, Taipei, Taiwan

REFERENCES:
- [Background] Aduen JF, Stapelfeldt WH, Johnson MM, Jolles HI, Grinton SF, Divertie GD, Burger CD. Clinical relevance of time of onset, duration, and type of pulmonary edema after liver transplantation. Liver Transpl. 2003 Jul;9(7):764-71. doi: 10.1053/jlts.2003.50103. PMID 12827567
- [Derived] Wu CY, Cheng YJ, Hung MH, Lin IJ, Sun WZ, Chan KC. Association between Early Acute Respiratory Distress Syndrome after Living-Donor Liver Transplantation and Perioperative Serum Biomarkers: The Role of Club Cell Protein 16. Biomed Res Int. 2019 Apr 11;2019:8958069. doi: 10.1155/2019/8958069. eCollection 2019. PMID 31111072